CLINICAL TRIAL: NCT02493387
Title: Should Elderly Patients With Atrial Fibrillation be Offered Physiotherapist Group Exercise or Can Physical Activity on Prescription (PAP) be Used as an Alternative
Brief Title: Supervised Exercise Compared to PAP in Patients With Permanent Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Goteborg Flimmer
Record Dates: First submitted 2015-07-06; First posted 2015-07-09 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Atrial Fibrillation
Keywords: Physiotherapist led group-based exercise; Physical activity; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise group (Experimental): The group-based exercise program consists of 60-minute sessions twice a week for 3 months, including central circulatory exercise performed on an ergometer cycle and muscle training, and one or two occasions of home-based exercise. The exercise program are designed after the patients requirements and with the intensity 13-17 on the RPE 6-20 scale
  Interventions: Other: Exercise
- PAP group (Active Comparator): The patients randomized PAP will receive a PAP prescription and a physical activity diary. The PAP and physical activity diary will be followed up at 6 and 12 weeks after the inclusion.
  Interventions: Other: Physical activity

INTERVENTIONS:
Other: Exercise — The group-based exercise program consists of 60-minute sessions twice a week for 3 months, including central circulatory exercise performed on an ergometer cycle and muscle training, and one or two occasions of home-based exercise. The exercise program are designed after the patients requirements and with the intensity 13-17 on the Borg RPE 6-20 scale
  Arms: Exercise group
Other: Physical activity — The patients randomized PAP will receive a PAP prescription and a physical activity diary. The PAP and physical activity diary will be followed up at 6 and 12 weeks after the inclusion.
  Arms: PAP group

SUMMARY:
Atrial fibrillation is the most common arrhythmia, and physical activity and exercise are sometimes avoided due to symptoms such as palpitations, fatigue and anxiety. Physiotherapist-led group based exercise as part of cardiac rehabilitation is rare for this group of patients, the method physical activity on prescription is used to encourage the patient to increase their physical activity level in order to reduce the risk of premature morbidity and mortality. However, mostly in this method you do not know the patient's ability to perform the prescribed amount of physical activity, and its effect on physical fitness has not been studied in patients with heart disease, neither has the effect of physiotherapist led group-based exercise in patients with atrial fibrillation. The aim was to investigate the impact of physiotherapy led group-based exercise compared to physical activity on prescription in patients with atrial fibrillation regarding the level of physical fitness, physical activity, heart rate and health related quality of life (HR-QoL).

DETAILED DESCRIPTION:
Ninety consecutive patients aged 65-85 years, visiting the cardiology clinic at Alingsås Hospital, Sahlgrenska University Hospital and primary care in the western part of Sweden will be asked to participate in the study. Inclusion criteria are permanent atrial fibrillation verified with electrocardiogram (ECG), left ventricular ejection fraction (EF) ≥ 45% and no significant valvular lesions verified by ultrasound. Exclusion criteria: Coronary event or angina pectoris within 3 months prior to inclusion, stroke with residual symptoms, presence of pacemaker or not able to participate in functional tests due to other disabilities, or to read Swedish. Physical fitness will be measured by a symptom limited bicycle test and a muscle endurance test. Physical activity will be measured by accelerometer and the International Physical Activity Questionnaire (IPAQ),HR-QoL will be measured by Short form (SF-36).

After the tests and return of accelerometer the patients will be randomized either to physiotherapist led group-based exercise or motivated interviewing and physical activity on prescription (PAP). The group-based exercise program consists of 60-minute sessions twice a week for 3 months, including central circulatory exercise performed on an ergometer cycle and muscle training, and two occasions of home-based exercise. The exercise program are designed after the patients requirements and with the intensity 13-17 on the Borg RPE 6-20 scale. The patients randomized to PAP will receive a PAP prescription and a physical activity diary. The PAP and physical activity diary will be followed up at 6 and 12 weeks after the inclusion. After three months all patients will perform the same tests as in baseline. A written informed consent will be obtained by the patients.

ELIGIBILITY:
Inclusion Criteria:

* permanent atrial fibrillation verified with electrocardiogram (ECG),
* left ventricular ejection fraction (EF) ≥ 45% and
* no significant valvular lesions verified by echocardiography

Exclusion Criteria:

* Coronary event or angina pectoris within 3 months prior to inclusion,
* stroke with residual symptoms,
* presence of pacemaker or
* not able to participate in functional tests due to other disabilities, or
* to read Swedish.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-01; Primary Completion 2018-06 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Physical fitness | 3 months
  Working capacity in watt

SECONDARY OUTCOMES:
Physical activity | 3 months
  Physical activity measured by accelerometer and questionnaire
Health related quality of life | 3 months
  questionnaire Short form SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Asa Cider, Phd RPT, Study Director — Institute of Neuroscience and Physiology/Physiotherapy
Locations (1):
- Sahlgrenska University Hospital and Alingsås Hospital, Gothenburg, Sweden